CLINICAL TRIAL: NCT06756958
Title: Reliability and Validity of Pittsburgh Rehabilitation Participation Scale During Robot Therapy Among Patients with Stroke
Brief Title: Reliability and Validity of Pittsburgh Rehabilitation Participation Scale During Robot Therapy
Status: Terminated | Type: Observational
Why Stopped: The researcher, who recruit, resigned.
Sponsor: National Rehabilitation Center, Seoul, Korea (Other Government)
Responsible Party: Principal Investigator, Kim, Jung Hwan, Team manager, National Rehabilitation Center, Seoul, Korea
Other Study IDs: NRC-2017-04-037
Record Dates: First submitted 2024-11-10; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Stroke
Keywords: participation; robot; scale; rehabilitation
MeSH Terms: conditions — Stroke | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention (observational study) — No intervention (observational study: The study participants were inpatient and were given robot-assisted gait training routinely.)

SUMMARY:
Reliability and validity of Pittsburgh Rehabilitation Participation Scale during robot therapy among patients with stroke

ELIGIBILITY:
Inclusion Criteria:

* patients with stroke or traumatic brain injury
* inpatient in rehabilitation center

Exclusion Criteria:

* brain tumor
* spinal cord injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those who participated the tethered-robot assisted gait training, had the history of brain lesion and adimitted in the rehabilitation center.
  Those who gave the informed consent about this study.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Rehabilitation Participation Scale | through study completion, an average of 3 year
  Pittsburgh Rehabilitation Participation Scale could be 1 (none), 2, 3, 4, 5, or 6 (excellent).
  Excellent (6): If the patient participated in all exercises or activities with maximal effort, finished all exercises or activities, and actively took interest in exercises or activities and/or future therapy sessions.
  None (1): patient refused entire session, or did not participate in any exercises or activities in session.
  In this study, a participant typically gets 12 sessions of robot assisted gait training. Just after the each session, Pittsburgh Rehabilitation Participation Scale is assigned as 1 to 6.
  For example, in a virtual case, the participant gets the score of 1, 1, 2, 2, 3, 3, 4, 4, 5, 5, 6, and 6 (median =3.5). the participant gets 12 numbers of outcome score and median of Pittsburgh Rehabilitation Participation Scale.

SECONDARY OUTCOMES:
modified Barthel Index | baseline and 4 weeks from baseline
  Modified Barthel Index measures basic activities of daily life. Lowest score is zero and means no function. Highiest score is 100, best function.
10m walk | baseline and 4 weeks from baseline
Borg scale | baseline and 4 weeks from baseline
  Borg scale measures perceived exertion during the test. It ranges 13 to 20. 13 means easy. 20 means hardest.
6 min walk | baseline and 4 weeks from baseline
motricity index | baseline and 4 weeks from baseline
Berg balance scale | baseline and 4 weeks from baseline
  Berg balance scale is the combination of 16 5-point-Likert-scale-like ordinal scale of 0 to 4.
  O means no balance. 56 means the maximal balance as the criteria.
Trunk impairment scale | baseline and 4 weeks from baseline
  Scores range from a minimum of 0 to a maximum of 23. Zero means no balance. 23 means maximal balance and trunk function.
Function in sitting test | baseline and 4 weeks from baseline
Modified Rankin Scale for Neurologic Disability | baseline and 4 weeks from baseline
  Modified Rankin Scale for Neurologic Disability could be 0, 1, 2, 3, 4, 5, or 6.
  Zero (0) means no negative symptoms et al as the criteria. 6 means means dead condition (death) as the criteria.
Functional Ambulatory Category | baseline and 4 weeks from baseline
Timed Timed Up and Go test | baseline and 4 weeks from baseline
Manual Muscle Testing | baseline and 4 weeks from baseline
modified Ashworth scale | baseline and 4 weeks from baseline
  Modified Ashworth scale could be 0, 1, 1+, 2, 3, or 4. Zero (0) means no spasticity as the criteria. 4 means means maximal spasticity as the criteria.
National Institutes of Health Stroke Scale | baseline and 4 weeks from baseline
  0 to 24 points. Zero (0) means no deficits as the criteria. 24 means means maximal deficits as the criteria.

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - National Rehabilitation Center, Seoul
  - Jung Hwan Kim, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Description site of the present study — http://nrc.go.kr